CLINICAL TRIAL: NCT04934423
Title: Analysis of Inflammatory Predictors and Differences in Gene Expression in Patients With Cognitive Impairment Responders and Non-responders to Neurostimulation: Clinical Trial, Double-Blind, Randomized
Brief Title: Analysis of Inflammatory Predictors and Gene Expression in Patients With Mild Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Suellen Marinho Andrade, Principal Researcher and Professor, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCL/Genes
Record Dates: First submitted 2021-02-09; First posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-02

CONDITIONS: Cognitive Decline
Keywords: Mild cognitive impairment; Direct Current Transcranial Stimulation; Inflammatory biomarkers; Gene expression
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled clinical trial will be conducted with patients diagnosed with Mild Cognitive Impairment, submitted to Direct Current Transcranial Stimulation sessions in a primary clinical trial. Both studies are in accordance with the guidelines of the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) (Moher & Chan, 2014), which is considered a tool composed of minimal contents of a clinical trial protocol.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study design in question involves patients with MCI, submitted to an intervention protocol, which includes: G1) active vs. G2) tDCS sham. These participants will be assessed previously for eligibility, then randomized to receive tDCS sham or active. All researchers responsible for the evaluation before and after the interventions will be blinded to the type of treatment the patient will receive (active stimulation or sham). The effectiveness of the masking mechanism will be assessed at the time of the last interview with patients when they will be asked about their opinion as to whether the electric current producing system was on or off.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tDCS (Experimental): tDCS active, for 30 minutes for 5 consecutive days, with an anode positioned in the left dorsolateral prefrontal cortex and cathode electrode placed over the right supraorbital area. The EEG International 10-20 system will be taken as a reference. The current intensity will be defined from computational modeling, using Nuclear Magnetic Resonance (MRI) to estimate and individualize a dose to be administered.
  Interventions: Device: Direct Current Transcranial Stimulation - tDCS
- Sham tDCS (Sham Comparator): The electrodes will be positioned in the same way as in the intervention group. However, individuals in this group will receive a stimulation that will last only 20-30 seconds. Subsequently, the device is switched off, no longer emitting current.
  Interventions: Device: Sham Intervention

INTERVENTIONS:
Device: Direct Current Transcranial Stimulation - tDCS — Active intervention
  Arms: active tDCS
Device: Sham Intervention — Direct Current Transcranial Stimulation - Sham intervention
  Arms: Sham tDCS

SUMMARY:
A randomized, double-blind, placebo-controlled clinical trial will be conducted, using data from participants who met the diagnostic criteria for mild cognitive impairment and who participated in a primary clinical trial that investigated the effectiveness of treatment with tDCS for patients with this pathology. The study in question seeks to investigate differences in inflammatory profile and gene expression in peripheral blood of patients with MCI responders and non-responders to treatment with tDCS, where it is intended to establish a profile of biomarkers that can predict disease progression. Primary study participants will be assessed previously for eligibility, then randomized to receive sham or active tDCS. Then, they will be invited to participate in the prediction analysis study to identify the inflammatory profile and gene expression. The participants' venous blood will be collected during the clinical examination on the first day of treatment, before the first session of tDCS, with a new collection after the last session, that is, at the baseline and the end point of our study.

DETAILED DESCRIPTION:
Healthy aging is associated with several changes in cortical function and these physiological differences are often interpreted as successful adaptation when cognitive performance is maintained; however, cognitive ability is not always preserved in aging. Mild cognitive impairment (MCI) is a cognitive decline syndrome commonly referred to as an intermediate phase between the expected cognitive decline of aging and pathological cognitive decline linked to dementia and generally does not interfere with daily activities. Pharmacological interventions have shown little positive impact and fail to demonstrate realizable benefits in mitigating cognitive decline in individuals with MCI and in preventing progression to Alzheimer's disease (AD). With this, there is a growing interest in exploring the benefits of non-pharmacological interventions such as Transcranial Direct Current Stimulation (tDCS), which can be a treatment modality to address the electrophysiological onset, deficits of metabolic and functional neural activation observed in MCI. Although tDCS has been studied in different dementias, there are still few studies investigating its use for MCI, with a significant lack of research in this area. Another issue to be explored is changes in the levels of biomarkers in body fluids and in specific brain regions of these patients, as they may allow the detection of cognitive changes even before the appearance of MCI. Different proteomic and genetic markers can result in a more accurate prediction of who will develop AD dementia in the future. The study in question seeks to investigate differences in the inflammatory profile and gene expression in the peripheral blood of patients with MCI responders and non-responders to treatment with tDCS, where it is intended to establish a profile of biomarkers that can predict the progression of the disease. Data from participants who met the diagnostic criteria for MCI and who participated in a clinical trial that investigated the effectiveness of treatment with tDCS for patients with this pathology will be used. Thus, it is necessary to mention the importance of early identification of the incipient forms of cognitive deficits, for the development of effective treatments. Several randomized controlled trials are underway to try to provide clinical evidence for the development of biomarkers that should provide the clinician with new tools to identify and treat MCI.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with CCL will be included
* Individuals of both sexes, aged 65 and over
* Individuals who do not have diagnosis of dementia

Exclusion Criteria:

* Subjects with unstable medical conditions
* Patients with metallic implants and pacemakers
* Epileptic patients
* Individuals using drugs / alcohol
* Those who are under regular use of hypnotics and benzodiazepines up to two weeks before the start of the study
* Those who are using medication with cholinergic inhibitors for more than two months before this clinical trial

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function | Evaluations will be carried out in the pre-intervention (T0)
  To assess the primary outcome, the Mini Mental State Examination (MMSE) or Mini-Mental State Examination (MMSE), developed in the United States and published in 1975, will be used, whose maximum score is 30 points and includes questions about memory, attention , orientation, language and visuospatial skills (Folstein, Folstein, & McHugh, 1975).
  We will adopt the 24-point score for the standard cut, following recommendations expressed in the literature (Anthony, Le Resche, Niaz, Von Korff, & Folstein, 1982; Folstein, Folstein, & McHugh, 1975). In order to avoid false positives and false negatives, we will perform the stratification by levels or years of schooling, as educational level is the main predictor of MMSE performance (Bertolucci, Brucki, Campacci, & Juliano, 1994).

SECONDARY OUTCOMES:
Inflammatory biomarkers | The assessment will be carried out at time T1 (baseline).
  We will analyze three inflammatory cytokines Il-6, Il-10 and tumor necrosis factor (TNFα) from a blood sample to compare their levels between the group treated with active current, responders and non-responders to neurostimulation.
Genetic Biomarkers | The assessment will be carried out at time T1 (baseline)
  For the genotyping of Neuregulin and alpha-synuclein markers, researchers will follow the method developed by Chomczynski and Sacchi (1987). Total RNA from peripheral blood sample will be extracted using Trizol reagent (Invitrogen). The results will be used as a prediction of the response to neurostimulation.